CLINICAL TRIAL: NCT06892431
Title: A Phase II Clinical Study of JMT101 Injection Combined With Mitoxantrone Liposome Injection in the Treatment of Patients With Recurrent or Metastatic Nasopharyngeal Cancer Who Have Failed At Least Two Prior Lines of Treatment
Brief Title: JMT101 Combined With Mitoxantrone Liposome for Nasopharyngeal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JMT101-019
Record Dates: First submitted 2025-03-21; First posted 2025-03-24 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Recurrent or Metastatic Nasopharyngeal Cancer; Patients Who Have Experienced Treatment Failure at Least Second-line Chemotherapy
MeSH Terms: conditions — Recurrence; Nasopharyngeal Neoplasms | interventions — Capecitabine; Docetaxel; Gemcitabine; Injections

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, positive-controlled Phase II
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JMT101 injection + Mitoxantrone Hydrochloride Liposome Injection; (Experimental): Treatment Group A: JMT101 Injection 6 mg/kg, intravenous drip, Q2W. Mitoxantrone Hydrochloride Liposome Injection 16 mg/m2, intravenous drip, Q4W.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome; Drug: JMT101 injection
- JMT101 + Mitoxantrone Liposome; (Experimental): Treatment Group B: JMT101 Injection 6 mg/kg, intravenous drip, Q2W. Mitoxantrone Hydrochloride Liposome Injection 20 mg/m2, intravenous drip, Q4W.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome; Drug: JMT101 injection
- Monotherapy chemotherapy regimens selected by the investigator. (Active Comparator): the dosage of capecitabine is 1000 mg/m2, taken orally twice daily, administered on D1-14 (Days 1-14) of each cycle, with every 3 weeks as one cycle (Q3W); the dosage of gemcitabine is 1000 mg/m2, administered via intravenous drip on D1 and D8 (Day 1 and Day 8) of each cycle, Q3W; the dosage of docetaxel is 75 mg/m2, administered via intravenous drip on D1 of each cycle, Q3W.
  Interventions: Drug: Capecitabine; Drug: Docetaxel injection; Drug: Gemcitabine hydrochloride for injection

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome — Mitoxantrone Hydrochloride Liposome Injection 20mg/m2, or 16mg/m2, intravenous drip, Q4W.
  Arms: JMT101 + Mitoxantrone Liposome;; JMT101 injection + Mitoxantrone Hydrochloride Liposome Injection;
Drug: JMT101 injection — JMT101 Injection 6 mg/kg, intravenous drip,
  Other Names: Recombinant Humanized Anti-Epidermal Growth Factor Receptor Monoclonal Antibody Injection
  Arms: JMT101 + Mitoxantrone Liposome;; JMT101 injection + Mitoxantrone Hydrochloride Liposome Injection;
Drug: Capecitabine — The dosage of capecitabine is 1000 mg/m2, taken orally twice daily, administered on D1-14 (Days 1-14) of each cycle, with every 3 weeks as one cycle (Q3W);
  Arms: Monotherapy chemotherapy regimens selected by the investigator.
Drug: Docetaxel injection — The dosage of docetaxel is 75 mg/m2, administered via intravenous drip on D1 of each cycle, Q3W.
  Arms: Monotherapy chemotherapy regimens selected by the investigator.
Drug: Gemcitabine hydrochloride for injection — The dosage of gemcitabine is 1000 mg/m2, administered via intravenous drip on D1 and D8 (Day 1 and Day 8) of each cycle, Q3W;
  Arms: Monotherapy chemotherapy regimens selected by the investigator.

SUMMARY:
This study is a randomized, open-label, multicenter Phase II clinical study, with the objective to assess the efficacy and safety of JMT101 Injection combined with Mitoxantrone Hydrochloride Liposome Injection in patients with recurrent/metastatic nasopharyngeal cancer who have failed at least two prior lines of treatment.

DETAILED DESCRIPTION:
Participants will be screened within 28 days prior to treatment, and those who meet the inclusion criteria and do not meet any of the exclusion criteria will be enrolled in this study. Enrolled participants will be randomly assigned in a 1:1:1 ratio to the following treatment groups, with each group planned to include 30-50 participants:

Mitoxantrone hydrochloride liposome will be administered for up to 6-8 cycles. After 6 cycles of administration, the investigator will decide whether to continue administration up to 8 cycles based on the patient's benefit-risk situation. JMT101 and the investigator-selected single-agent chemotherapy regimen will continue to be administered until progressive disease (PD) as assessed by the investigator according to RECIST v1.1 criteria, intolerable toxicity, withdrawal of informed consent by the subject, initiation of new anti-tumor treatment, loss to follow-up, death, or the end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign the written ICF;
2. Aged 18-75 years old (inclusive), male or female;
3. Patients with nasopharyngeal cancer who have experienced treatment failure after prior PD-(L)-1 inhibitor therapy and at least second-line chemotherapy (including at least one line containing platinum);
4. According to RECIST v1.1, there is at least one measurable lesion, and the lesion has not previously undergone radiotherapy or has shown definite progression after radiotherapy;
5. ECOG PS score of 0-1;
6. Estimated lifespan of at least 3 months;
7. Have adequate organ function, laboratory test meets the following criteria (has not received transfusion or hematopoietic stimulating factor treatment within 14 days):(1)Hematology: a. Absolute neutrophil count ≥1.5×109/L; b. Platelet count ≥100×109/L; c. Hemoglobin ≥90 g/L.(2)Liver function: a. Total bilirubin ≤1.0×ULN; for participants with metastases to liver, total bilirubin ≤1.5×ULN; b. Alanine aminotransferase and aspartate aminotransferase ≤1.5×ULN, for participants with metastases to liver, alanine aminotransferase and aspartate aminotransferase ≤2.5×ULN. (3)Renal function: Creatinine ≤1.5×ULN; or creatinine clearance ≥50 mL/min (calculated according to the Cockcroft-Gault formula).(4)Coagulation function: International normalized ratio (INR) ≤ 1.5×ULN; activated partial thromboplastin time (APTT) ≤ 1.5×ULN;
8. Women of childbearing potential must use highly effective contraception.

Exclusion Criteria:

1. Previously received EGFR monoclonal antibody therapy for recurrent/metastatic nasopharyngeal cancer;
2. Have previously received treatment with doxorubicin or other anthracyclines, and the cumulative dose of doxorubicin exceeds 350 mg/m2 (Equivalent dose calculation for anthracyclines: 1 mg doxorubicin = 2 mg epirubicin = 2 mg daunorubicin = 0.5 mg idarubicin = 0.45 mg mitoxantrone);
3. History of drug allergy to the active or inactive excipients of any study drug, or to drugs with similar chemical structure or class as these two drugs;
4. Have received anti-tumor treatments within 2 weeks prior to the first dose of study drug, including hormone therapy, biological therapy, immunization therapy, local perfusion of anti-tumor drugs, or traditional Chinese medicines and/or Chinese patent drugs indicated for the treatment of nasopharyngeal cancer;
5. Have received local radiotherapy (including radionuclide therapy such as strontium-89) within 2 weeks prior to the first dose of study drug; have received irradiation of more than 30% of bone marrow or have received wide-field radiotherapy within 4 weeks prior to randomization;
6. Uncontrolled serous cavity effusions requiring frequent drainage or medical intervention within 14 days prior to the first dose;
7. Have undergone major surgery or had severe traumatic injury within 4 weeks prior to the first dose of study drug, or it is expected to undergo major surgery during the study period. Some clinical procedures such as vascular access placement and aspiration biopsy are allowed;
8. Currently receiving long-term immunosuppression therapy (e.g., cyclosporine) or have other diseases requiring treatment with systemic corticosteroids (i.e., prednisone over 10 mg/day or other corticosteroids at equivalent physiological doses), excluding those receiving local glucocorticoid therapy via nasal spray, inhalation, or other routes;
9. Participants with metastases to meninges or spinal cord compression; participants with symptomatic and/or unstable brain metastasis, unless the participant has completed definitive treatment and has been stable for at least 2 weeks prior to randomization without the need for steroid therapy. Participants with asymptomatic brain metastases may be enrolled if the investigator assesses that there is no indication for immediate curative treatment;
10. Subjects who have taken strong CYP3A4 inducers or inhibitors within 2 weeks prior to the first dose of study drug, or who cannot suspend the use of strong CYP3A4 inducers and inhibitors during the study;
11. Participants with a history of autoimmune diseases, a history of immunodeficiency, including positive for HIV, or other acquired or immunodeficiency congenital diseases, or a history of organ transplant;
12. Presence of active infection (e.g., the subject is receiving anti-infection therapy), including uncontrolled active hepatitis b, active hepatitis c, active syphilis, active tuberculosis, etc.; Patients with a history of human hepatitis B virus (HBV) infection may be considered for enrollment if they meet all of the following criteria: a. Have no co-infection with hepatitis C virus (HCV) and no history of HCV infection; b. Participants with active HBV infection may also be enrolled if they can receive at least 2 weeks of antiviral therapy before starting study treatment, and after treatment their HBV DNA is less than 100 IU/mL and transaminases are less than 1×ULN.
13. Severe or uncontrolled cardiovascular disorder requiring treatment, including but not limited to
14. Refractory nausea, vomiting, chronic gastrointestinal disease, inability to swallow drugs orally, or previous subtotal small bowel resection, etc., and have conditions that seriously affect gastrointestinal absorption as judged by the investigator.
15. Prior to initiating treatment, have not yet adequately recovered (i.e., to ≤ Grade 1, excluding hypodynamia or alopecia) from toxicities and/or complications caused by any interventions;
16. Participants with other malignant tumors currently or with a history of other active malignant tumors within 5 years prior to the first study treatment (except for clinically cured localized tumors;
17. History of interstitial lung disease (ILD), history of drug-induced ILD, history of radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD;
18. Women who are pregnant or breastfeeding;
19. The researchers believe that the subjects are not suitable to participate in this clinical study due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) per RECIST v1.1 | Up to approximately 30 months after the first participant is enrolled

SECONDARY OUTCOMES:
Disease control rate (DCR) per RECIST 1.1 | Up to approximately 30 months after the first participant is enrolled
Duration of response (DoR) per RECIST 1.1 | Up to approximately 30 months after the first participant is enrolled
Progression free survival (PFS) per RECIST 1.1 | Up to approximately 30 months after the first participant is enrolled
Overall survival(OS) | Up to approximately 30 months after the first participant is enrolled
Frequency and severity of AEs (NCI CTCAE 5.0) | Up to approximately 30 months after the first participant is enrolled
The plasma concentrations of JMT101, total mitoxantrone, and free mitoxantrone | Up to approximately 15 months after the first participant is enrolled
The incidence of JMT101 anti-drug antibodies (ADAs), titers, and neutralizing antibodies (NAbs, if applicable) | Up to approximately 15 months after the first participant is enrolled
The correlation between EGFR expression level and efficacy | Up to approximately 15 months after the first participant is enrolled

IPD SHARING:
Plan to Share IPD: No